CLINICAL TRIAL: NCT01065506
Title: Smoking Termination Enhancement Project (STEP)
Acronym: STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southern Methodist University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jasper Smits, Ph.D., Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA027533 (NIH); 1R01DA027533-01 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices; Health Promotion; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care plus Wellness Program (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Treatment; Drug: Nicotine Patch; Behavioral: Wellness Program
- Standard Care plus Exercise Program (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Treatment; Drug: Nicotine Patch; Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment — Cognitive Behavioral Treatment
Drug: Nicotine Patch — Nicotine Patch
Behavioral: Wellness Program — Wellness Program
  Arms: Standard Care plus Wellness Program
Behavioral: Aerobic Exercise — Aerobic Exercise
  Arms: Standard Care plus Exercise Program

SUMMARY:
The primary aim of this research study (STEP) is to compare the effectiveness of two smoking cessation programs that integrate counseling and nicotine replacement with either a wellness program or exercise. This will help us to determine whether different lifestyle interventions (wellness or exercise) help increase the effectiveness of current standard programs for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years old
2. Capable of providing informed consent, attend all study visits and comply with the protocol
3. Daily smoker for at least one year and currently smoke an average of at least 10 cigarettes per day
4. Report a motivation to quit smoking in the next month of at least 5 on a 10-point scale
5. Score of 20 or greater on 16-item Anxiety Sensitivity Index
6. Physically inactive as defined as participating in moderate-intensity exercise less than 2 days/week (duration must be 30 minutes or less each time)

Exclusion Criteria:

1. Use of other tobacco products
2. General medical condition(s) that contraindicate exercise
3. Resting blood pressure of ≥ 160 systolic and/or 100 diastolic who are not receiving treatment for high blood pressure
4. Blood lipid levels ≥ 240 mg/dl with LDL-C ≥ 160 mg/dl or triglyceride levels ≥ 300 mg/dl (individuals receiving medical treatment for lipid abnormalities with lipid levels above the cut-offs will be eligible with physician written approval)
5. Body mass index ≥40
6. Currently suicidal or high suicide risk
7. Current or past psychotic disorders of any type, or comorbid psychiatric conditions that are relative or absolute contraindications to the use of any treatment option in the study protocol
8. Currently pregnant, planning on becoming pregnant in the next year, or current breastfeeding
9. Alcohol or drug dependence; abuse of depressants, dissociative anesthetics, hallucinogens, opioids, or cocaine within the last 6 months
10. Psychotherapy initiated within the past three months, or ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety or mood disorder other than general supportive therapy
11. Current use of any psychotherapy or pharmacotherapy for smoking cessation not provided by the researchers, including Chantix, Zyban, Welbutrin and Nortriptyline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, PhD, Principal Investigator — Southern Methodist University; Michael Zvolensky, PhD, Principal Investigator — University of Houston
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

REFERENCES:
- [Background] Tart CD, Leyro TM, Richter A, Zvolensky MJ, Rosenfield D, Smits JA. Negative affect as a mediator of the relationship between vigorous-intensity exercise and smoking. Addict Behav. 2010 Jun;35(6):580-5. doi: 10.1016/j.addbeh.2010.01.009. Epub 2010 Feb 1. PMID 20171786
- [Background] Smits JA, Rosenfield D, Mather AA, Tart CD, Henriksen C, Sareen J. Psychotropic medication use mediates the relationship between mood and anxiety disorders and obesity: findings from a nationally representative sample. J Psychiatr Res. 2010 Nov;44(15):1010-6. doi: 10.1016/j.jpsychires.2010.04.007. PMID 20434171
- [Background] Medina JL, Vujanovic AA, Smits JA, Irons JG, Zvolensky MJ, Bonn-Miller MO. Exercise and coping-oriented alcohol use among a trauma-exposed sample. Addict Behav. 2011 Mar;36(3):274-7. doi: 10.1016/j.addbeh.2010.11.008. Epub 2010 Nov 10. PMID 21111538
- [Background] Smits JA, Bonn-Miller MO, Tart CD, Irons JG, Zvolensky MJ. Anxiety sensitivity as a mediator of the relationship between moderate-intensity exercise and coping-oriented marijuana use motives. Am J Addict. 2011 Mar-Apr;20(2):113-9. doi: 10.1111/j.1521-0391.2010.00115.x. Epub 2011 Feb 1. PMID 21314753
- [Background] Smits JA, Tart CD, Rosenfield D, Zvolensky MJ. The interplay between physical activity and anxiety sensitivity in fearful responding to carbon dioxide challenge. Psychosom Med. 2011 Jul-Aug;73(6):498-503. doi: 10.1097/PSY.0b013e3182223b28. Epub 2011 Jun 23. PMID 21700713
- [Background] Mathew AR, Norton PJ, Zvolensky MJ, Buckner JD, Smits JA. Smoking Behavior and Alcohol Consumption in Individuals With Panic Attacks. J Cogn Psychother. 2011 Feb 1;25(1):61-70. doi: 10.1891/0889-8391.25.1.61. PMID 21915160
- [Background] Zvolensky MJ, Buckner JD, Norton PJ, Smits JA. Anxiety, Substance Use, and Their Co-Occurrence: Advances in Clinical Science. J Cogn Psychother. 2011;25(1):3-6. doi: 10.1891/0889-8391.25.1.3. PMID 21857769
- [Background] Deboer LB, Tart CD, Presnell KE, Powers MB, Baldwin AS, Smits JA. Physical activity as a moderator of the association between anxiety sensitivity and binge eating. Eat Behav. 2012 Aug;13(3):194-201. doi: 10.1016/j.eatbeh.2012.01.009. Epub 2012 Jan 28. PMID 22664396
- [Derived] Smits JA, Zvolensky MJ, Davis ML, Rosenfield D, Marcus BH, Church TS, Powers MB, Frierson GM, Otto MW, Hopkins LB, Brown RA, Baird SO. The Efficacy of Vigorous-Intensity Exercise as an Aid to Smoking Cessation in Adults With High Anxiety Sensitivity: A Randomized Controlled Trial. Psychosom Med. 2016 Apr;78(3):354-64. doi: 10.1097/PSY.0000000000000264. PMID 26513517
- [Derived] Smits JA, Zvolensky MJ, Rosenfield D, Marcus BH, Church TS, Frierson GM, Powers MB, Otto MW, Davis ML, DeBoer LB, Briceno NF. The efficacy of vigorous-intensity exercise as an aid to smoking cessation in adults with elevated anxiety sensitivity: study protocol for a randomized controlled trial. Trials. 2012 Nov 13;13:207. doi: 10.1186/1745-6215-13-207. PMID 23148822

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 150 enrolled participants, 7 participants completed a baseline assessment, then subsequently dropped out of the study before receiving any treatment. 7 participants were used as pilots. Accordingly, results are reported for the remaining 136 participants.
Groups:
- Standard Care Plus Wellness Program: Cognitive Behavioral Treatment: Cognitive Behavioral Treatment
  Nicotine Patch: Nicotine Patch
  Wellness Program: Wellness Program consisting of thrice weekly sessions involving discussion of various wellness topics (e.g., diet, sun care, cancer prevention) and generating small wellness-related goals
- Standard Care Plus Exercise Program: Cognitive Behavioral Treatment: Cognitive Behavioral Treatment
  Nicotine Patch: Nicotine Patch
  Aerobic Exercise: Aerobic Exercise thrice weekly (on a treadmill)
Period: Overall Study
Arm/Group | Standard Care Plus Wellness Program | Standard Care Plus Exercise Program
Started | 64 | 72
End of Treatment | 44 | 37
4-Month Follow-Up | 35 | 34
Completed | 32 | 34
Not Completed | 32 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care Plus Wellness Program | Standard Care Plus Exercise Program | Total
Number analyzed (Participants) | 64 | 72 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.39 (11.30) | 43.12 (11.26) | 44.19 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 28 | 36 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 18 | 28
  White | 49 | 51 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 64 | 72 | 136
ASI-3 [Mean (Standard Deviation); unit: units on a scale] — Throughout treatment and follow-up, we assessed Anxiety Sensitivity using the Anxiety Sensitivity Index-3 (ASI-3). Recent research has supported using a cut-off score of 23 to identify high AS individuals with this instrument. ASI was assessed via self-report online prior to each assessment visit. ASI scores range from 0 to 72. Lower anxiety sensitivity scores in this study are indicative of better outcomes.
  units on a scale | 18.63 (10.36) | 18.04 (12.72) | 18.32 (11.62)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Abstained From Smoking at 10 and 30 Weeks Post Quit Day
Description: Point Prevalence Abstinence (PPA) was defined as not smoking [even a single puff] at the end of treatment and/or on the day of follow-up
Time Frame: End of treatment (10 weeks post quit day) and 30-week follow-up
Population: Participants who completed the end of treatment assessment
Measure: Number; unit: number of participants
Arm/Group | Standard Care Plus Wellness Program | Standard Care Plus Exercise Program
Number analyzed (Participants) | 44 | 37
number of participants
  End of treatment | 5 | 9
  Follow-up (n=35, 34) | 4 | 9

ADVERSE EVENTS:
Arm/Group | Standard Care Plus Wellness Program | Standard Care Plus Exercise Program
Serious Adverse Events (participants affected / at risk) | 1/64 | 1/72
Other Adverse Events (participants affected / at risk) | 0/64 | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care Plus Wellness Program (N=64) | Standard Care Plus Exercise Program (N=72)
Malignant melanoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vertebrae fractures (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not obtained during study sessions; deemed unrelated to study procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No